CLINICAL TRIAL: NCT05512650
Title: Use of Virtual Reality for Musculoskeletal Pain
Brief Title: Virtual Reality and Meditation for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Brigham and Women's Hospital (Other); Rheumatology Research Foundation (Other)
Responsible Party: Principal Investigator, Nancy Baker, Chair of and Associate Professor in Department of Occupational Therapy, Tufts University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021P001499
Record Dates: First submitted 2022-08-12; First posted 2022-08-23 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Virtual Reality; Meditation; Pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- VR first (Active Comparator): At their first visit, subjects will engage in a virtual reality meditation while wearing the VR headset. At their second visit, they will engage in a non-immersive meditation without the 3D VR aspect.
  Interventions: Device: Virtual Reality Meditation; Device: Non-VR Meditation
- VR second (Active Comparator): At their first visit, subjects will engage in a non-immersive meditation without the 3D VR aspect. At their second visit, they will engage in a virtual reality meditation while wearing the VR headset.
  Interventions: Device: Virtual Reality Meditation; Device: Non-VR Meditation

INTERVENTIONS:
Device: Virtual Reality Meditation — Participants will be set up in the VR equipment. They will engage and follow along with a 10-20 minute guided meditation through the VR. The meditation program may include simulated movement, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
Device: Non-VR Meditation — Participants will engage and follow along with a 10-20 minute guided meditation on a computer screen placed before them. The meditation program may include simulated movement visuals, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.

SUMMARY:
Fibromyalgia (FM) is a particularly debilitating rheumatological syndrome which affects millions of adults in the United States. The condition presents with widespread chronic muscular pain and reduced pain thresholds, fatigue, insomnia, and negative affect. Chronic pain that is caused by FM can have significant effects on physical function, psychological parameters, and overall quality of life. Currently, there is a need for safe and effective non-pharmacologic pain-management strategies for FM, and research has shown that virtual reality (VR) may be a useful tool for some of these clients. The literature has suggested improvements in pain scores on a visual analog scale (VAS) for adults with a variety of rheumatological issues, including FM. Additional research has demonstrated that affect was improved for clients with FM who participated in a 10-minute VR mindfulness session. Such findings highlight the potential benefits of VR and mindfulness meditation for clients with FM. However, there is a great deal that remains unknown about the effectiveness of these pain management techniques. Therefore, this pilot study will examine and compare the effectiveness of combining VR and meditation for improving symptoms of FM in adults. We hypothesize that a VR meditation session will facilitate greater improvements in pain, affect, and physiological vital stats as compared to a non-immersive meditation intervention.

DETAILED DESCRIPTION:
Current treatments for fibromyalgia (FM) include pharmaceutical pain medications (ranging from over the counter to prescription opioids) as well as psychological programs with components of relaxation, cognitive therapy, and activity management. However, pain medications are not fully effective, can be addictive, and can cause hyperalgesia, and there is little research on psychological interventions for FM.

One treatment that has demonstrated some efficacy for reducing chronic pain is meditation. Various studies have demonstrated that there are generally reductions in affective pain for those who practice meditation. Another promising treatment option for FM is virtual reality (VR). VR is an immersive 3D experience during which the participant wears a headset or helmet which simulates the sensation of being elsewhere. There is evidence which shows that VR can be an effective treatment for pain reduction. However, most studies which utilize VR as a method of pain reduction focus on acute pain and studies looking at VR for chronic pain are scarce.

One preliminary study examined the utility of VR in treating FM. Results from this study showed that positive affect increased after participants engaged in a 10-minute meditation and mindfulness VR session. Further, they found a slight reduction in the negative impact of FM on overall life and wellbeing, as measured by the FM Impact Questionnaire (FIQ). However, small sample sizes and the addition of other adjunctive therapies limit the significance of these study results. Additional research on VR and meditation for the treatment of FM and other rheumatological conditions also demonstrated reductions in pain scores, offering promising data on meditation and VR being used in combination.

Given the promising literature on VR and meditation, this study will aim to further the field of knowledge surrounding use of VR meditation for reducing pain and increasing affect for adults with FM. Despite the encouraging data on using these interventions for FM, it is unknown whether the immersive aspect of the VR is helping to improve results. This pilot study will aim to address this question by comparing an immersive VR meditation session with a non-immersive, typical meditation for FM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18 and older (no upper limit)
2. Diagnosis of fibromyalgia with a minimum average pain level of 3 over the last week
3. English-speaking
4. Willing and able to visit the Brigham and Women's Pain Management Center site on two separate occasions to participate in the study

Exclusion Criteria:

1. Unwilling to put on VR headset
2. Experience a seizure in the last 5 years
3. Cognitive impairment
4. Hearing/visual deficit
5. Active, contagious skin infection
6. Eye infections
7. Has a pacemaker or defibrillator
8. Has a hearing aid
9. History of myocardial infarction or other serious cardiovascular condition
10. Current peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Baker, Principal Investigator — Tufts University
Locations (1):
- Brigham and Women's Pain Management Center, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venuturupalli RS, Chu T, Vicari M, Kumar A, Fortune N, Spielberg B. Virtual Reality-Based Biofeedback and Guided Meditation in Rheumatology: A Pilot Study. ACR Open Rheumatol. 2019 Nov 11;1(10):667-675. doi: 10.1002/acr2.11092. eCollection 2019 Dec. PMID 31872189
- [Background] Botella C, Garcia-Palacios A, Vizcaino Y, Herrero R, Banos RM, Belmonte MA. Virtual reality in the treatment of fibromyalgia: a pilot study. Cyberpsychol Behav Soc Netw. 2013 Mar;16(3):215-23. doi: 10.1089/cyber.2012.1572. PMID 23496678
- [Background] Ahmadpour N, Randall H, Choksi H, Gao A, Vaughan C, Poronnik P. Virtual Reality interventions for acute and chronic pain management. Int J Biochem Cell Biol. 2019 Sep;114:105568. doi: 10.1016/j.biocel.2019.105568. Epub 2019 Jul 12. PMID 31306747
- [Background] Herrero R, Garcia-Palacios A, Castilla D, Molinari G, Botella C. Virtual reality for the induction of positive emotions in the treatment of fibromyalgia: a pilot study over acceptability, satisfaction, and the effect of virtual reality on mood. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):379-84. doi: 10.1089/cyber.2014.0052. PMID 24892201
- [Background] Hennard J. A protocol and pilot study for managing fibromyalgia with yoga and meditation. Int J Yoga Therap. 2011;(21):109-21. PMID 22398352
- [Background] Ngian GS, Guymer EK, Littlejohn GO. The use of opioids in fibromyalgia. Int J Rheum Dis. 2011 Feb;14(1):6-11. doi: 10.1111/j.1756-185X.2010.01567.x. Epub 2010 Aug 23. PMID 21303476
- See also: Centers for Disease Control (CDC) on Fibromyalgia — https://www.cdc.gov/arthritis/fibromyalgia/?CDC_AAref_Val=https://www.cdc.gov/arthritis/types/fibromyalgia.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Reality Meditation 1st/Non Virtual Reality Meditation 2nd: Virtual Reality Meditation: Participants will be set up in the VR equipment. They will engage and follow along with a 10-20 minute guided meditation through the VR. The meditation program may include simulated movement, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
  Non Virtual Reality Meditation: Non-VR Meditation: Participants will engage and follow along with a 10-20 minute guided meditation on a computer screen placed before them. The meditation program may include simulated movement visuals, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
- Non Virtual Reality Meditation 1st/Virtual Reality Meditation 2nd: Non-VR Meditation: Participants will engage and follow along with a 10-20 minute guided meditation on a computer screen placed before them. The meditation program may include simulated movement visuals, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
  Virtual Reality Meditation: Participants will be set up in the VR equipment. They will engage and follow along with a 10-20 minute guided meditation through the VR. The meditation program may include simulated movement, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
Period: Overall Study
Arm/Group | Virtual Reality Meditation 1st/Non Virtual Reality Meditation 2nd | Non Virtual Reality Meditation 1st/Virtual Reality Meditation 2nd
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Virtual Reality Meditation 1st/ NonVr 2nd: Virtual Reality Meditation: Participants will be set up in the VR equipment. They will engage and follow along with a 10-20 minute guided meditation through the VR. The meditation program may include simulated movement, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
  Non-VR Meditation: Participants will engage and follow along with a 10-20 minute guided meditation on a computer screen placed before them. The meditation program may include simulated movement visuals, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
- Non Virtual Reality Meditation 1st/VR Meditaiton 2nd: Non-VR Meditation: Participants will engage and follow along with a 10-20 minute guided meditation on a computer screen placed before them. The meditation program may include simulated movement visuals, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
  Virtual Reality Meditation: Participants will be set up in the VR equipment. They will engage and follow along with a 10-20 minute guided meditation through the VR. The meditation program may include simulated movement, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Meditation 1st/ NonVr 2nd | Non Virtual Reality Meditation 1st/VR Meditaiton 2nd | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Pain Numerical Rating Scale [NRS] (Change From Pre-intervention to Post-intervention)
Description: Measures the intensity of pain on an 11-point scale, ranging from 0-10. 0 is "no pain", and 10 is "pain as bad as you can imagine".
Time Frame: 20 minutes after the 10 minute intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Non Virtual REality Medition: Non-VR Meditation: Participants will engage and follow along with a 10-20 minute guided meditation on a computer screen placed before them. The meditation program may include simulated movement visuals, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
Arm/Group | Virtual Reality Meditation | Non Virtual REality Medition
Number analyzed (Participants) | 9 | 9
score on a scale | 4.4 (1.7) | 4.8 (1.8)

2. Secondary Outcome: Positive and Negative Affect Scale [PANAS]
Description: This twenty-item self-report questionnaire measures the extent to which the participant felt various emotions right now. There are two scales, positive affect and negative affect. This questionnaire uses a 5-point Likert scale, from 1 (very slightly or not at all) to 5 (extremely). This questionnaire will assess the participant's psychological state. There are 10 items for each scale ad each scale is summed seperately from the items to form a Positive Affect outcome and a Negative Affect scale. The total for each of these scales is 10 to 50. A higher score indicated more of that affect so a high score on the Positive Affect is considered better while a lower score on the Negative Affect is considered better.
Time Frame: 20 minutes post the 10 minute meditation intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Non Virtual Reality Meditation: Non-VR Meditation: Participants will engage and follow along with a 10-20 minute guided meditation on a computer screen placed before them. The meditation program may include simulated movement visuals, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
Arm/Group | Virtual Reality Meditation | Non Virtual Reality Meditation
Number analyzed (Participants) | 9 | 9
score on a scale
  Panas Postivie | 25.8 (9.1) | 27.3 (8.4)
  Panas Negative | 10.7 (.9) | 11.3 (2.3)

3. Secondary Outcome: Quantitative Sensory Testing (QST) - Pain Threshold
Description: Measurements of pain thresholds for bilateral trapezius muscles using a pressure algometer which is a fsmall force guage that can apply controlled pressure to specific points on the body. The algometer quantifies the minimum pressure required to induce pain. It is applied to specific muscles and the tester gradually increases the pressure on that muscle belly until the participant reports that the pressure is painful. For our study we applied pressure to the trapezious muscle Pain Threshold is measured in pounds per square inch and the range is from 0 to infinity. A higher score is considered to be a more positive outcome (e.g. the person is tolerating more pressure before identifying it is painful)
Time Frame: 20 minutes post the 10 minute meditation intervention
Measure: Mean (Standard Deviation); unit: pounds per square inch
Groups:
- VR Meditation: Virtual Reality Meditation: Participants will be set up in the VR equipment. They will engage and follow along with a 10-20 minute guided meditation through the VR. The meditation program may include simulated movement, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
- Non VR Meditation: Non-VR Meditation: Participants will engage and follow along with a 10-20 minute guided meditation on a computer screen placed before them. The meditation program may include simulated movement visuals, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
Arm/Group | VR Meditation | Non VR Meditation
Number analyzed (Participants) | 9 | 9
pounds per square inch | 1.6 (.9) | 1.8 (1.4)

4. Secondary Outcome: Blood Pressure
Description: We obtained Systolic and Diastolic blood pressure using an automated BP cuff. We converted these two scores into a single called the Mean Arterial Pressure which is the average pressure in a person's arteries during one cardiac cycle. The equation used is 1/3(SBP)+2/3(DBP). Thus, this outcome is turned into a single value for analysis. A lower score is considered a better scores.
Time Frame: Immediately after a 10 minute meditation intervention
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | VR Meditation | Non VR Meditation
Number analyzed (Participants) | 9 | 9
mm Hg | 82.6 (15.1) | 81.5 (12.3)

5. Secondary Outcome: Heart Rate
Description: Heart rate was obtained using an automated BP cuff. The scale is beats per minute with a range of 50 to ~200 beats per minute. A lower score is a more positive score
Time Frame: Immediately after a 10 minute meditation intervention
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | VR Meditation | Non VR Meditation
Number analyzed (Participants) | 9 | 9
Beats per minute | 75.7 (11.2) | 75.2 (11.2)

6. Secondary Outcome: Quantitative Sensory Testing (QST) - Temporal Summation
Description: Temporal summation involves touching the participants finger multiple times with a precisely calibrated sharp object and asking for their rating of the discomfort experienced from the touch using the NRS. The NRS measures the intensity of pain on an 11-point scale, ranging from 0-10. 0 is "no pain", and 10 is "pain as bad as you can imagine". A lower score is considered a more positive outcome
Time Frame: 20 minutes post the 10 minute meditation intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Meditation | Non VR Meditation
Number analyzed (Participants) | 9 | 9
score on a scale | 1.8 (1.3) | 1.6 (1.5)

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | VR Meditation | Non VR Meditation
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
Small Sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT05512650/Prot_002.pdf